CLINICAL TRIAL: NCT05997524
Title: Clinical Efficacy of Trastuzumab in Combination With Capecitabine and Oxaliplatin for the Treatment of HER2-positive Advanced Gastric Cancer: A Multicenter, Phase II Study
Brief Title: Clinical Efficacy of Trastuzumab in Combination With Capecitabine and Oxaliplatin for the Treatment of HER2-positive Advanced Gastric Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Ishtiaq-Ur-Rahim, Principal Investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHL/2021/01
Record Dates: First submitted 2023-08-06; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Advanced Gastric Carcinoma
MeSH Terms: interventions — Trastuzumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tras-Capox (Experimental)
  Interventions: Drug: Trastuzumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab was administered at a loading dose of 8 mg/kg followed by 6 mg/kg infusion every 3 weeks (q3w).
Drug: Oxaliplatin — Oxaliplatin was administrated as a 130 mg/m2 infusion, q3w, for up to 6 cycles.
Drug: Capecitabine — Capecitabine 1000 mg/m2 was given orally twice daily on days 1-14 followed by a 7-day rest interval.

SUMMARY:
Trastuzumab plus chemotherapy prolonged the median overall survival in patients with human epidermal growth factor receptor 2 (HER2)-positive advanced gastric cancer (AGC). Among chemotherapy regimens, oxaliplatin is generally more convenient and tolerable than cisplatin, and becoming an increasingly popular option for the treatment of AGC. The aim of the study was to evaluate the efficacy and safety of trastuzumab in combination with capecitabine and oxaliplatin (CAPOX) in HER2-positive AGC.

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive AGC defined as either HER2 immunohistochemistry (IHC) 3+ or IHC 2+ and fluorescence in situ hybridization (FISH)+ with no history of previous treatment.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Loco-regional and Distant Tumor Control After Completion of Treatment | 12 months
  Response Evaluation Criteria in Solid Tumors was used to measure outcome:
  Complete response (CR): Disappearance of all target lesions. Partial response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Progressive disease (PD): At least a 20% increase in the sum of diameters of target lesions.
  Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 28 months
Overall survival (OS) | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarwar Alam, MBBS, Mphil, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No